CLINICAL TRIAL: NCT04248816
Title: Increasing Surveillance Rates for Hepatocellular Carcinoma Among Cirrhotic Patients
Brief Title: Hepatocellular Carcinoma Surveillance in Cirrhotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shivan J Mehta, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 834574; 5P30AG03456-10 (Other Grant/Funding Number: National Institute on Aging)
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis
Keywords: Behavioral Economics; Screening; Outreach
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Experimental): Standard of care
  Interventions: Behavioral: Usual care
- Opt-out (Experimental): Facilitated outreach and opt-out framing
  Interventions: Behavioral: Opt-out
- Opt-out + Incentive (Experimental): Facilitated outreach and opt-out framing plus a financial incentive
  Interventions: Behavioral: Opt-out + Incentive

INTERVENTIONS:
Behavioral: Usual care — Subjects will receive outreach through their providers as is standard of care.
  Arms: Usual Care
Behavioral: Opt-out — Research staff will send a letter to patients encouraging them to get a surveillance ultrasound and include an order slip for them to get it done at a health system facility.
  Arms: Opt-out
Behavioral: Opt-out + Incentive — Research staff will send a letter to patients encouraging them to get a surveillance ultrasound and include an order slip plus an unconditional $20 incentive for them to get it done at a health system facility.
  Arms: Opt-out + Incentive

SUMMARY:
This is a 3-arm pilot randomized controlled trial applying behavioral economic approaches (opt-out framing and financial incentives) to encourage patients with liver cirrhosis to complete regular surveillance ultrasounds which may allow for earlier diagnosis of and better outcomes for hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
There is a substantial burden of HCC-related morbidity and mortality: The age-adjusted incidence rates of HCC have tripled in the US since the 1980s due to the burden of hepatitis C virus (HCV) and the epidemic of non-alcoholic fatty liver disease (NAFLD). The overwhelming majority of HCC in the US occurs in the setting of cirrhosis. Early diagnosis of HCC dictates survival: The American Association for the Study of Liver Diseases (AASLD) recommends biannual HCC surveillance for all patients with cirrhosis using an abdominal ultrasound. These guidelines seek to maximize early diagnosis of HCC which leads to earlier detection and improved survival because early-stage HCC is curable, with 70% 5-year survival compared to 5% in advanced disease.

HCC surveillance rates are suboptimal: Despite longstanding published guidelines for HCC surveillance, adherence is low, with surveillance rates ranging from 15-30% in the US. Two RCTs have tested interventions to increase HCC surveillance, including electronic reminders for primary care providers and mailed reminders (with or without navigators), but neither has been scalable, produced durable responses, or increased surveillance rates above 50%.

This is a 3-arm pilot randomized controlled trial applying behavioral economic approaches (opt-out framing and financial incentives) to encourage patients with liver cirrhosis to complete regular surveillance ultrasounds which may allow for earlier diagnosis of and better outcomes for hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18+ years old
* Current diagnosis of cirrhosis or advanced fibrosis
* 1 or more visits to a Penn Gastroenterology/Hepatology practice in the preceding two years
* Currently followed by Penn Gastroenterology/Hepatology
* Must live in the Philadelphia Metropolitan Statistical Area

Exclusion Criteria:

* History of HCC or other liver carcinoma diagnosis
* History of liver transplant
* Completed HCC screening within the past 7 months
* Have a future screening scheduled
* Have a different screening modality recommended by their physician (MRI, CT, etc.)
* Patients with metastatic cancer
* Patients receiving hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Opt-out | Opt-out + Incentive
Started | 123 | 245 | 247
Completed | 116 | 224 | 222
Not Completed | 7 | 21 | 25
Not completed — Ineligible post-randomization | 7 | 21 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Opt-out | Opt-out + Incentive | Total
Number analyzed (Participants) | 116 | 224 | 222 | 562
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (11.6) | 61.4 (10.9) | 62.9 (11.0) | 62.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 101 | 92 | 243
  Male | 66 | 123 | 130 | 319
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 11 | 26
  Not Hispanic or Latino | 106 | 213 | 207 | 526
  Unknown or Not Reported | 2 | 4 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 9 | 15 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 46 | 88 | 94 | 228
  White | 66 | 116 | 104 | 286
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 11 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: HCC Screening Completion
Description: The percentage of subjects who have a surveillance abdominal ultrasound.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Usual Care | Opt-out | Opt-out + Incentive
Number analyzed (Participants) | 116 | 224 | 222
Percentage of participants | 27.6 [19.5 to 35.7] | 54.5 [47.9 to 61.0] | 54.1 [47.5 to 60.6]

2. Secondary Outcome: HCC Screening Method
Description: The percentage of subjects who have any hepatocellular carcinoma surveillance.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Usual Care | Opt-out | Opt-out + Incentive
Number analyzed (Participants) | 116 | 224 | 222
Percentage of patients | 32.8 [24.2 to 41.3] | 59.4 [52.9 to 65.8] | 57.2 [50.7 to 63.7]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were not monitored or assessed as the intervention involves receiving a gift card and/or a letter by mail. Receiving mail has few risks and is unlikely to cause serious adverse events. No drug, medical device or medical procedure was under investigation.
Arm/Group | Usual Care | Opt-out | Opt-out + Incentive
All-Cause Mortality (participants affected / at risk) | 2/123 | 6/245 | 12/247
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT04248816/Prot_SAP_000.pdf